CLINICAL TRIAL: NCT05183178
Title: Switching From Ticagrelor to Prasugrel in Patients With Acute Coronary Syndrome-a Stepped Wedge Cluster Randomized Evaluation in the SWEDEHEART-registry
Brief Title: Switching From Ticagrelor to Prasugrel in Patients With Acute Coronary Syndrome
Acronym: SWITCH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Region Skane (Other); Region Halland (Other); Region Gävleborg (Other); Region Örebro County (Other); Region Västerbotten (Other Government); Jämtland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWITCH v 1.0 2020-12-10
Record Dates: First submitted 2021-11-19; First posted 2022-01-10 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized evaluation in the SWEDEHEART-registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor (Active Comparator): Current standard of care
  Interventions: Drug: Ticagrelor 90 mg
- Prasugrel (Experimental): New standard of care
  Interventions: Drug: Prasugrel 10 mg p.o

INTERVENTIONS:
Drug: Prasugrel 10 mg p.o — Prasugrel 10 mg once daily p.o. Patient >75 years of age or <60 kg will receive 5 mg prasugrel OD.
  Arms: Prasugrel
Drug: Ticagrelor 90 mg — Ticagrelor 90 mg twice daily p.o.
  Arms: Ticagrelor

SUMMARY:
This study proposes to conduct the switch from ticagrelor to prasugrel in an organized stepwise manner, to allow for the evaluation of the relative efficacy of prasugrel versus ticagrelor using a stepped-wedge cluster randomized trial design.

DETAILED DESCRIPTION:
The SWITCH SWEDEHEART trial is a prospective, multicenter, open-label, cross-sectional, stepped wedge cluster randomized clinical study, in which administrative regions in Sweden will constitute the clusters. Many administrative regions have already decided to switch from ticagrelor to prasugrel for the treatment of patients with ACS. The order in which the regions make the switch will be randomly assigned. At the start of the study, all regions will utilize and prescribe ticagrelor as the P2Y12 inhibitor drug of choice for patients with ACS. After 9 months, one cluster will switch from ticagrelor to prasugrel as the P2Y12 inhibitor of choice for patients with ACS. Every 9 months, an additional cluster will switch to prasugrel until all clusters have switched from ticagrelor to prasugrel. Study enrollment will be stop 9 months after the last cluster has switched to prasugrel. The study will be terminated when 1-year follow-up has been concluded for all patients.

All patients who are hospitalized due to acute coronary syndrome in any of the health care regions over the course of the study period will be included. All patients will be treated according to local treatment guidelines at the time of the index hospitalization (prasugrel or ticagrelor) for at least 12 months. Patients with relative or absolute contra-indications for the study drugs or patients experiencing side effects requiring treatment changes will be treated according to current guidelines at the discretion of the treating physician.

The patients will be identified via the Swedish Web-System for Enhancement and Development of Evidence-Based Care in Heart Disease Evaluated According to Recommended Therapies (SWEDEHEART) registry. The events at 1 year will be identified and extracted from Patient registry (Socialstyrelsen), Population registry (Folkbokföringen), Causes of death registry (Socialstyrelsen). Compliance with the treatment after the transition from ticagrelor to prasugrel will be followed through Dispensed drug registry (Socialstyrelsen).

Primary objective:

• To investigate the clinical efficacy of Prasugrel compared to Ticagrelor for the treatment of patients hospitalized for acute coronary syndrome

Secondary objectives:

* To investigate the cost effectiveness of Prasugrel compared to Ticagrelor for the treatment of patients hospitalized for acute coronary syndrome (ICD-10 codes: I21-I22), with respect to the 1-year outcomes.
* To investigate clinical safety of Prasugrel compared to Ticagrelor for the treatment of patients hospitalized for acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for Acute coronary syndrome, as defined by the European Society of Cardiology, at any hospital participating in the study, and included in the SWEDEHEART registry during index hospitalization
* Age ≥ 18 years.

Exclusion Criteria:

* Patients on oral anticoagulation therapy
* Previous stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative risk (%) | 1-year
  Cumulative risk of death, myocardial infarction or stroke

SECONDARY OUTCOMES:
Cost effectiveness ratio (%) | 1-year
  Cost effectiveness of Prasugrel compared to Ticagrelor.
Bleeding or Death ratio (%) | Within 30 days
  Bleeding or death (in-hospital) within30 days

OTHER OUTCOMES:
Cumulative incidence of death (%) | 1-year
  Risk of death
Cumulative incidence myocardial infarction or death (%) | 1-year
  Risk of myocardial infarction or death
The composite of all-cause death, myocardial infarction, or stroke (%) | Within 30 days
  The composite of all-cause death, myocardial infarction, or stroke
Cumulative incidence of major bleeding (%) | Within 30 days
  Major bleeding
The composite of all-cause death, myocardial infarction, stroke or urgent revascularization (%) | Within 30 days
  The composite of all-cause death, myocardial infarction, stroke or urgent revascularization (defined as re-intervention due to acute coronary syndrome)
The cumulative incidence of endpoints (%) | Within 30 days and 1 year
  The cumulative incidence of the following endpoints;
  * All-cause mortality
  * Definite or probable stent thrombosis
  * Definite stent thrombosis
  * Myocardial infarction
  * Stroke
  * Major bleeding
  * Ischemia-driven target vessel revascularization
  * Ischemia-driven revascularization
  * Interruption of study drug within 1 year
  * Interruption of dual antiplatelet therapy within 1 year
Cumulative all-cause mortality (%) | 2 years and yearly up to 15 years.
  Cumulative all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Elmir Omerovic, MD, PhD, Principal Investigator — Sahlgrenska Universitetssjukhus
Locations (1):
- Dep. Cardiology, Skånes universitetssjukhus, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided